CLINICAL TRIAL: NCT06734468
Title: Personalized Approach to Promote Healthy Aging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Susan Racette, Professor, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00020392
Record Dates: First submitted 2024-12-08; First posted 2024-12-16 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-10

CONDITIONS: Aging; Aging, Healthy
Keywords: Healthy aging; Aging; Healthspan
MeSH Terms: interventions — Nutritional Status; Sleep; Exercise

STUDY DESIGN:
Intervention Model Description: A pre-post design will be used, with all participants receiving the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lifestyle Intervention (Experimental): All participants will receive an intervention.
  Interventions: Behavioral: Lifestyle Management

INTERVENTIONS:
Behavioral: Lifestyle Management — Each subject will receive a personalized intervention plan, comprised of:
  1. An individualized exercise plan guided by a mobile phone app.
  2. Healthy diet and nutrition recommendations.
  3. Theriome metabolomics testing and individualized recommendations that include dietary supplements.
  4. Guidance on healthy sleep patterns, stress management, and maximizing social engagement, as appropriate.
  Other Names: Nutrition; Sleep habits; Stress management; Social engagement; Exercise

SUMMARY:
The goal of this clinical trial study is to evaluate the impact of a personalized lifestyle intervention on improving healthspan. The primary questions of interest are whether the personalized intervention will result in improvements in muscle function, immune function, and cognitive function in adults aged 50-85 years. Participants will complete baseline assessments, receive an individualized intervention plan for approximately 3 months, and then complete post-intervention assessments. The intervention includes an exercise plan, nutrition recommendations, and general lifestyle goals that will be personalized to each participant.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 years of age
* Non-smoking
* Ambulatory without the need of an assistive device (walker, cane, etc.) and able to perform exercise testing and exercise training
* English speaking
* Owns a smart phone

Exclusion Criteria:

* Minors and adults younger than age 50 years and older than 85 years
* Pregnant women
* Adults who are unable to provide informed consent
* Prisoners

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
VO2 max | From baseline to the end of the intervention at 3 months.
  A maximal treadmill exercise test with respiratory gas exchange analysis to assess cardiorespiratory fitness.
Biodex | From baseline to the end of the intervention at 3 months.
  A Biodex will be used to assess leg muscle power and strength.

SECONDARY OUTCOMES:
World Health Organization Quality of Life Survey | From baseline to the end of the intervention at 3 months.
  We will assess quality of life with the WHO_QoL. The WHO_QoL is scored from 0-100 with a higher score indicating a higher quality of life.
Pittsburgh Sleep Quality Index | From baseline to the end of the intervention at 3 months.
  This questionnaire assesses sleep quality. The PSQI is scored on a scale from 0-21 with a higher score indicating higher sleep quality.
Handgrip strength | From baseline to the end of the intervention at 3 months.
  A hand-held dynamometer will be used to measure handgrip strength.
Dual Energy X-ray Absorptiometry (DXA) | From baseline to the end of the intervention at 3 months.
  A DXA scan will be used to assess body composition and bone mineral density.
Waist circumference | From baseline to the end of the intervention at 3 months.
  Waist circumference will be measured at the superior border of the iliac crest.
Hip circumference | From baseline to the end of the intervention at 3 months.
  Hip circumference will be measured at the maximal protrusion of the buttocks.
Systolic blood pressure | From baseline to the end of the intervention at 3 months.
  Systolic blood pressure will be measured at rest.
Diastolic blood pressure | From baseline to the end of the intervention at 3 months.
  Diastolic blood pressure will be measured at rest.
Digit Symbol Substitution Test (DSST) | From baseline to the end of the intervention at 3 months.
  The DSST assesses cognition and cognitive impairment.
Montreal Cognitive Assessment (MoCA) | From baseline to the end of the intervention at 3 months.
  The MoCA assesses cognition and cognitive impairment. The MoCA is scored out of 30 points and a higher score indicates better cognitive function.
Short Physical Performance Battery | From baseline to the end of the intervention at 3 months.
  A performance test to assess balance and physical function.
Low Density Lipoprotein Cholesterol | From baseline to the end of the intervention at 3 months.
  A test assessing calculated LDL cholesterol.
Hemoglobin A1C Concentration | From baseline to the end of the intervention at 3 months.
  This will assess a participants HbA1C.
Insulin Concentration | From baseline to the end of the intervention at 3 months.
  This test will assess a participants fasting insulin.
Geriatric Depression Scale (GDS) | From baseline to the end of the intervention at 3 months.
  This survey assesses feelings of depression in older adults. The GDS is scored from 0-15, with a higher score indicating more feelings of depression.
Generalized Anxiety Disorder (GAD)-7 | From baseline to the end of the intervention at 3 months.
  This survey assess feelings of anxiety. The GAD-7 is scored from 0-21, with higher scores indicating higher feelings of anxiety.
Perceived Stress Scale | From baseline to the end of the intervention at 3 months.
  This survey assesses perceived stress. This survey is scored from 0-40 with higher scores indicating higher stress.
High Density Lipoprotein Cholesterol | From baseline to the end of the intervention at 3 months.
  A blood test measuring HDL cholesterol.
Brief Resilience Scale | From baseline to the end of the intervention at 3 months.
  This survey assess a participants resilience. This survey is scored from 0-30 with higher scores indicating a higher level of resilience.
Non-High Density Lipoprotein Cholesterol | From baseline to the end of the intervention at 3 months.
  A blood test measuring non-HDL cholesterol.
Very Low Density Lipoprotein Cholesterol | From baseline to the end of the intervention at 3 months.
  A blood test measuring VLDL cholesterol.
CD3 T cells | From baseline to the end of the intervention at 3 months.
  This test will measure how many CD3 Mature T Cells are in the blood. This will be reported as a percentage.
CD4 T cells | From baseline to the end of the intervention at 3 months.
  This test will measure the CD4 T cells in the blood. This will be reported as a percentage.
CD8 T cells | From baseline to the end of the intervention at 3 months.
  This test will measure the CD8 T cells in the blood. This will be reported as a percentage.
Natural Killer cells | From baseline to the end of the intervention at 3 months.
  This test will measure the NK cells in the blood. This will be reported as a percentage.
B cells | From baseline to the end of the intervention at 3 months.
  This test will measure the B cells in the blood. This will be reported as a percentage.

OTHER OUTCOMES:
Resting metabolic rate | From baseline to the end of the intervention at 3 months.
  A test to assess how many calories the body burns at rest. RMR will be measured in the fasted state while the participant is supine.
Red Blood Cells | From baseline to the end of the intervention at 3 months.
  This will assess the number of red blood cells.
White blood cells | From baseline to the end of the intervention at 3 months.
  This will assess the number of white blood cells.
Platelets | From baseline to the end of the intervention at 3 months.
  This will assess the number of platelets in the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Wexford Innovation Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary outcomes will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available after all data have been collected, entered into the REDCap database, data cleaning procedures have been completed, and the primary articles have been published. Data will be available on or before 1/1/2028 and will remain available for a minimum of 3 years.
Access Criteria: The Arizona State University Research Data Repository can be accessed freely by investigators. This data repository has supporting information about the protocol and contact information for the investigative team.
URL: https://dataverse.asu.edu/